CLINICAL TRIAL: NCT06081582
Title: Toripalimab in Combination With Cetuximab，Cisplatin and 5-FU for Conversion Therapy of Locally Nonresectable Oral Cavity Squamous Cell Carcinoma （OCSCC）
Brief Title: Toripalimab in Combined With Cetuximab，Chemotherapy for Conversion Therapy of Locally Nonresectable OCSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yulong Zheng, Chief Physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220085C-R1
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab; Cetuximab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus Cetuximab，chemotherapy group (Experimental): All subjects received 2-cycle conversion therapy with the PD-1 inhibitor toripalimab combined with cetuximab, cisplatin, and 5-FU
  The dosage of medication used is as follows:
  Toripalimab: 240mg, Day1, Q3W；Cisplatin: 25mg/m2, Day1-3, Q3W；5-FU: 1000mg/m2, Day1-3, Q3W Cetuximab Day 1, 8, 15, Q3W, 400 mg/m2 initial dose; Afterwards, 250 mg/m2 per week
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — This study was conducted on 30 patients with initially unresectable locally advanced head and neck squamous cell carcinoma who underwent two cycles of PD-1 antibody (trepril monoclonal antibody) combined with fluorouracil, cisplatin, and cetuximab conversion therapy. The feasibility of radical surgery should be evaluated before surgical treatment.Three patients were enrolled in the safe induction period before the study began.
  The dosage of medication used is as follows:
  Toripalimab: 240mg, Day1, Q3W
  Cisplatin: 25mg/m2, Day1-3, Q3W（every 3 weeks）
  5-FU: 1000mg/m2, Day1-3, Q3W
  Cetuximab Day 1, 8, 15, Q3W, 400 mg/m2 initial dose; Afterwards, 250 mg/m2 per week
  Other Names: Drug: Cetuximab; Drug: Cisplatin; Drug: 5-FU

SUMMARY:
This is a prospective, single center phase II clinical study with a planned enrollment of 33 patients. The main objective is to evaluate the efficacy and safety of the PD-1 inhibitor toripalimab combined with cetuximab, cisplatin, and 5-FU regimen in the treatment of locally advanced oral squamous cell carcinoma patients who are initially unresectable.

DETAILED DESCRIPTION:
In the past decade, the treatment plan for non-surgical locally advanced HNSCC patients who are suitable for receiving synchronous radiotherapy and chemotherapy has remained unchanged, and innovative treatment methods are urgently needed. Based on the above research, immunotherapy combined with chemotherapy and immunotherapy combined with cetuximab have good efficacy and safety in non-surgical HNSCC patients. Therefore, combining PD-L1 antibodies with chemotherapy, surgery to further improve the efficacy of comprehensive treatment may become a new direction in tumor treatment. The achievement of pCR or MPR in conversion therapy is related to better OS and DFS outcomes in patients. In the era of immunotherapy, conversion therapy centered around surgery has become a hot topic in the field of treatment for locally advanced oral squamous cell carcinoma that cannot be surgically removed upon initial diagnosis.

There is no particularly preferred standard conversion chemotherapy regimen for patients with locally advanced head and neck squamous cell carcinoma that cannot be surgically removed initially. The combination of PD-1 inhibitor toripalimab, cetuximab, and chemotherapy may benefit the efficacy of these patients. Therefore, this prospective phase II clinical trial was designed to evaluate the efficacy and safety of PD-1 inhibitor toripalimab combined with chemotherapy and cetuximab conversion therapy in locally advanced oral squamous cell carcinoma patients who were initially unresectable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of tongue, floor of mouth, gingival, buccal
* Initial NCCN TNM stage III and IVA patients
* PS score 0-1 points
* Age≥18 years old
* Measurable lesions that meet RECIST 1.1 standards
* Normal function of important organs
* All patients must provide tissue specimens

Exclusion Criteria:

* Active, known or suspected autoimmune disease patients
* According to the judgment of the researcher, there are accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study by the patients
* Merge with other malignant tumors
* Subjects with known central nervous system metastasis and/or cancerous meningitis
* Uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage
* Received significant surgical treatment or obvious traumatic injury within the first 28 days of randomization
* Have experienced arterial/venous thrombotic events within the first 6 months of randomization, such as cerebrovascular accidents
* Individuals with a history of abuse of psychotropic substances who are unable to quit or have mental disorders
* Subjects with any severe and/or uncontrollable diseases
* Exclusion criteria related to concomitant medications
* Participated in other clinical trials within four weeks
* Have received preventive or attenuated vaccines within 4 weeks before the first administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Major pathological response（MPR） | through study completion; an average of 1 year
  To determine the major pathological response rate, defined as <10% viable tumor in the resection specimen, after two cycles of neoadjuvant Toripalimab Plus Cetuximab，Cisplatin and 5-FU in patients with Nonresectable Oral Cavity Squamous Cell Carcinoma （OCSCC）

CONTACTS AND LOCATIONS:
Overall Officials: Yulong Zheng, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Medical Onocology, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No